CLINICAL TRIAL: NCT01934504
Title: Defining Immune Tolerance in ANCA-associated Vasculitis (AAV)
Acronym: AAV
Status: Terminated | Type: Observational
Why Stopped: Slow accrual
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Other Study IDs: DAIT ITN051AI; AVATARS (Other: Immune Tolerance Network)
Record Dates: First submitted 2013-08-29; First posted 2013-09-04 (Estimated); Results first posted 2016-05-20 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-04

CONDITIONS: ANCA-Associated Vasculitis
Keywords: clinical tolerance; biomarker(s) identification
MeSH Terms: conditions — Anti-Neutrophil Cytoplasmic Antibody-Associated Vasculitis | interventions — Phlebotomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * peripheral blood mononuclear cells (PBMCs)
  * whole blood RNA
  * serum
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Tolerant AAV: Tolerant participants with AAV
  Interventions: Procedure: Venipuncture for blood sample collection
- Non-Tolerant AAV: Non-Tolerant participants with ANCA-associated vasculitis (AAV)
  Interventions: Procedure: Venipuncture for blood sample collection
- Healthy Controls: Healthy participants that fulfill eligibility criteria -similar in age to Tolerant and Non-Tolerant AAV participants.
  Interventions: Procedure: Venipuncture for blood sample collection
- AAV Discontinuing Immunosuppression: Participants have been in clinical remission and on minimal maintenance therapy for at least 2 years prior to screening. Their primary physicians have planned to discontinue immunosuppression medication in the next year after screening.
  Interventions: Procedure: Venipuncture for blood sample collection

INTERVENTIONS:
Procedure: Venipuncture for blood sample collection — Analysis samples from the blood sample collection at specific time points.
  Other Names: Peripheral venous blood draw

SUMMARY:
The goal of the study is to find biological markers (certain proteins or cellular markers found in a blood test) that will inform doctors which patients diagnosed with ANCA-associated vasculitis (AAV) are most likely to be able to stop their medications suppressing their immune systems and remain in remission.

DETAILED DESCRIPTION:
Anti-neutrophil cytoplasmic antibody (ANCA)-associated vasculitides (AAV) are small vessel vasculitides that typically follow a chronic course and are associated with serious illness and death.Three clinical conditions are recognized: microscopic polyangiitis (MPA); granulomatosis with polyangiitis (Wegener's, GPA); and eosinophilic granulomatosis with polyangiitis (EPA, formerly Churg Strauss Syndrome). Though these conditions have different clinical features, they can have overlapping immunological characteristics.

The precise cause of AAV is not understood, but there are clear genetic associations which, in the context of predisposing environmental factors, such as infections, may lead to development of disease. There are no diagnostic criteria for AAV, but there are validated classification criteria and disease definitions.

There is a need to find biological markers that define immunological tolerance so that immunotherapy medicines may be correctly changed and safely withdrawn in some people.

ELIGIBILITY:
Inclusion Criteria:

Tolerant AAV participants:

* Age 18 years or older
* Diagnosis of granulomatosis with polyangiitis (Wegener's, GPA) or microscopic polyangiitis (MPA) according to the definitions of the Chapel Hill Consensus Conference (CHCC)
* History of being myeloperoxidase (MPO)-ANCA positive during a disease flare
* In clinical remission with Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) = 0 and off all immunosuppression for ≥ 2 years
* Negative MPO-ANCA and proteinase 3 (PR3)-ANCA by ELISA at screening
* For women of child-bearing potential, a negative urine or serum pregnancy test at the time of screening
* Ability to sign and understand informed consent
* Willingness to comply with study procedures.

Non-Tolerant AAV participants:

* Age 18 years or older
* Diagnosis of granulomatosis with polyangiitis (Wegener's), GPA or microscopic polyangiitis (MPA) according to the definitions of the CHCC
* History of being MPO-ANCA positive during a disease flare
* Within the past 5 years, must have had a disease exacerbation, defined as an increase in the BVAS/WG score and re-institution of immunosuppressive therapy after therapy had been reduced or completely discontinued
* In clinical remission with BVAS/WG = 0 and on minimal maintenance therapy for ≥3 months prior to the screening visit. Minimal maintenance therapy is defined as:

  * Low-dose glucocorticoids (≤10 mg of prednisone or prednisolone daily) and/or:

    * Azathioprine ≤ 150mg daily or
    * Mycophenolate mofetil (MMF) ≤ 1 gram daily or mycophenolate sodium ≤ 720 mg daily.
* Positive MPO-ANCA by ELISA on at least 2 occasions within the last 52 weeks, the most recent result being within 8 weeks of visit -1
* For women of child-bearing potential, a negative urine or serum pregnancy test at the time of screening
* Ability to sign and understand informed consent
* Willingness to comply with study procedures.

Healthy Controls:

* Healthy participant age ≥18 years
* For women of child-bearing potential, a negative urine or serum pregnancy test at the time of screening
* Ability to sign and understand informed consent
* Willingness to comply with study procedures.

Exclusion Criteria:

Tolerant AAV Participants:

* Use of systemic intravenous (IV) or oral glucocorticoids for ˃ 1 month for any non-vasculitis indication within 8 weeks of the screening visit
* Any prior treatment with rituximab
* Presence of known chronic viral infections or autoimmune diseases
* History of malignancy, excluding non-melanomatous skin cancers or cervical cancer carcinoma in situ within 5 years of the screening visit.

Non-Tolerant AAV participants:

* Use of IV pulse glucocorticoids (methylprednisolone or other) or cyclophosphamide within the year prior to the screening visit
* Use of IV or oral glucocorticoids for > 1 month for any non- vasculitis indication within 8 weeks of screening visit
* Any prior treatment with rituximab
* Maintenance therapy with methotrexate within 3 months of the screening visit
* Presence of known chronic viral infections or other autoimmune diseases
* History of malignancy, excluding non-melanoma skin cancers or cervical cancer carcinoma in situ within 5 years of the screening visit.

Healthy Controls:

* Use of IV or oral glucocorticoids for > 1 month for any non-vasculitis indication within 8 weeks of the screening visit
* Presence of known chronic viral infections or other autoimmune diseases
* History of malignancy, excluding non-melanoma skin cancers or cervical cancer carcinoma in situ within 5 years of the screening visit.

AAV Participants Discontinuing Immunosuppression:

* Any prior treatment with rituximab
* Maintenance therapy with methotrexate within 3 months of the screening visit
* Presence of known chronic viral infections or other autoimmune diseases
* History of malignancy, excluding non-melanoma skin cancers or cervical cancer carcinoma in situ, within 5 years of the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Non-tolerant: Patients who have persistently active disease. Tolerant: Those patients who have become ANCA negative, having been ANCA positive at the time of their acute presentation but have been in prolonged disease- free remission off all immunotherapy for at least two years. Healthy controls: Individuals with similar age distribution to participants in the Non-tolerant and Tolerant cohorts.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2013-12; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Salama, MD, Study Chair — University College London, Centre for Nephrology
Locations (3):
- United Kingdom (3):
  - Addenbrooke's Hospital, Cambridge, England
  - University College London, Centre for Nephrology, London, England
  - Hammersmith Hospital, London, England

REFERENCES:
- See also: The National Institute of Allergy and Infectious Diseases — http://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with granulomatosis with polyangiitis (Wegener's, GPA) or microscopic polyangiitis, and a history positive for the presence of MPO-ANCA+ during disease flares were recruited for 3 cohorts; healthy participants were recruited for 1 cohort. Participants were recruited from 3 sites in Great Britain from Dec 2013 to Feb 2015.
Groups:
- Tolerant AAV: Subjects in the Tolerant ANCA-associated vasculitis (AAV) cohort have been in clinical remission with Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) scores of zero and have been off all immunosuppression medications for at least 2 years prior to screening. Subjects have blood samples and other assessments collected for analysis at Week 0 and Week 26.
- Non-Tolerant AAV: Subjects in the Non-Tolerant ANCA-associated vasculitis (AAV) cohort have had a disease exacerbation and re-institution of immunosuppressive therapy in the past 5 years. Subjects have also been in clinical remission with Birmingham Vasculitis Activity Score for Wegener's Granulomatosis (BVAS/WG) scores of zero and on minimal maintenance therapy for at least 3 months prior to screening. Subjects have blood samples and other assessments collected for analysis at Week 0 and Week 26.
- Healthy Controls: Healthy participants without autoimmune disease. Subjects have blood samples and other assessments collected for analysis at Week 0 and Week 26.
- AAV Discontinuing Immunosuppression: Subjects in the ANCA-associated vasculitis (AAV) Discontinuing Immunosuppression group have been in clinical remission with Birmingham Vasculitis Activity Score for Wegener's Granulomatosis BVAS/WG) scores of zero and on minimal maintenance therapy for at least 2 years prior to screening. The subjects' primary physicians have planned to discontinue immunosuppression medication in the next year after screening. Subjects have blood samples and other assessments collected for analysis at Week 0 and at 8 weeks after discontinuation of immunosuppression medication.
Period: Overall Study
Arm/Group | Tolerant AAV | Non-Tolerant AAV | Healthy Controls | AAV Discontinuing Immunosuppression
Started | 6 | 3 | 16 | 8
Completed | 5 | 3 | 11 | 1
Not Completed | 1 | 0 | 5 | 7
Not completed — Protocol Deviation | 0 | 0 | 0 | 2
Not completed — Study Terminated by Sponsor | 1 | 0 | 5 | 5

BASELINE CHARACTERISTICS:
Population: The baseline analysis population is defined as all participants who have undergone the Week 0 blood sample collection
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolerant AAV | Non-Tolerant AAV | Healthy Controls | AAV Discontinuing Immunosuppression | Total
Number analyzed (Participants) | 6 | 3 | 16 | 8 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 4 | 3 | 10
  >=65 years | 5 | 1 | 12 | 5 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.7 (13.5) | 58.3 (7.6) | 69.4 (7.1) | 64.8 (7.5) | 68.1 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 9 | 5 | 18
  Male | 4 | 1 | 7 | 3 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 3 | 16 | 8 | 33
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 2
  White | 5 | 3 | 15 | 6 | 29
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 6 | 3 | 16 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Tolerance Biomarker Identification
Description: Identification of biomarkers associated with clinical tolerance in patients with ANCA-associated vasculitis by comparative immunophenotyping of individual leukocyte subsets from tolerant and non-tolerant patients with AAV.
  Due to early study termination, data was not available to evaluate this endpoint.
Time Frame: Difference from baseline to week 26
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | Tolerant AAV | Non-Tolerant AAV | Healthy Controls | AAV Discontinuing Immunosuppression
Number analyzed (Participants) | 0 | 0 | 0 | 0

2. Secondary Outcome: Tolerance Signature Stability
Description: Measurement of the stability of a tolerance immune signature in patients with AAV over time.
  Due to early study termination, data was not available to evaluate this endpoint.
Time Frame: Baseline to Week 26
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | Tolerant AAV | Non-Tolerant AAV | Healthy Controls | AAV Discontinuing Immunosuppression
Number analyzed (Participants) | 0 | 0 | 0 | 0

3. Secondary Outcome: Tolerance Signature Versus Clinical Status
Description: Correlation of possible changes in the tolerance signature with changes in clinical status.
  Due to early study termination, data was not available to evaluate this endpoint.
Time Frame: Baseline to Week 26
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | Tolerant AAV | Non-Tolerant AAV | Healthy Controls | AAV Discontinuing Immunosuppression
Number analyzed (Participants) | 0 | 0 | 0 | 0

4. Secondary Outcome: Immunosuppression Associated Signature
Description: Definition of an immune signature associated with maintenance immunosuppression.
  Due to early study termination, data was not available to evaluate this endpoint.
Time Frame: Baseline to 8 Weeks Post-Immunosuppression Withdrawal
Population: No analyses were performed due to slow enrollment and early study closure.
Arm/Group | Tolerant AAV | Non-Tolerant AAV | Healthy Controls | AAV Discontinuing Immunosuppression
Number analyzed (Participants) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Subjects in Tolerant AAV, Non-Tolerant AAV, Healthy Controls were followed though Week 26. Subjects in Discontinuation group were followed until 8 weeks after discontinuing immunosuppression meds anytime between Week 0 and 52, for a max time of 60 weeks
Arm/Group | Tolerant AAV | Non-Tolerant AAV | Healthy Controls | AAV Discontinuing Immunosuppression
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/16 | 0/8
Other Adverse Events (participants affected / at risk) | 0/6 | 0/3 | 0/16 | 0/8

LIMITATIONS AND CAVEATS:
Study termination due to slow enrollment, resulting in no outcome analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No